CLINICAL TRIAL: NCT02751606
Title: Nano MRI on 7 Tesla: a Technical Validation Study in Rectal and Breast Cancer
Brief Title: Nano MRI on 7 Tesla in Rectal and Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7TNANO1
Record Dates: First submitted 2014-11-28; First posted 2016-04-26 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2017-09

CONDITIONS: Rectal Neoplasms; Breast Neoplasms
Keywords: Ferumoxtran; MRI Scans
MeSH Terms: conditions — Rectal Neoplasms; Breast Neoplasms | interventions — ferumoxtran-10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breast and rectal cancer (Experimental): Subjects will receive intravenous dose of ferumoxtran-10. 24-36 hours later a 7 Tesla MRI scan will be performed, to detect lymph node metastases. In rectal cancer patients the mesorectum will be imaged and for breast cancer patients this will be performed in the ipsilateral axilla. Subjects will also undergo a 3 Tesla MRI scan as a comparison to the 7 Tesla MRI scan.
  Interventions: Drug: ferumoxtran-10; Device: 7 Tesla MRI; Device: 3 Tesla MRI

INTERVENTIONS:
Drug: ferumoxtran-10 — ferumoxtran-10 will be administered intravenously one day prior to the MRI scan
Device: 7 Tesla MRI — Subjects undergo a 7 Tesla MRI scan
Device: 3 Tesla MRI — Subjects undergo a 3 Tesla MRI scan

SUMMARY:
This study evaluates the diagnostic accuracy of an USPIO contrast agent (ferumoxtran-10) in combination with 7 Tesla MRI to detect lymph node metastases in rectal and breast cancer.

DETAILED DESCRIPTION:
The Presence of lymph node metastases in cancer is a key factor for determining prognosis and forming an adequate treatment plan. Determining lymph node status, however, is a challenge. Ferumoxtran-10, an ultrasmall superparamagnetic iron oxide (USPIO) particle has proven to be a valuable contrast agent for detecting lymph node metastases using magnetic resonance imaging (MRI) in various types of cancer (also called nano-MRI). For small lymph node metastases (<5mm) the diagnostic accuracy of this technique does, however, drop substantially. Most of the studies that have been performed with these particles used a 1.5 Tesla or 3 Tesla MRI scanner. The investigators would like to increase the resolution of nano-MRI by using a 7 Tesla scanner, such that the investigators can increase the sensitivity of this technique for small lymph nodes. With this study the investigators would like to validate the results of this technique with pathology in rectal and breast cancer. In these cancer types many patients undergo a surgical lymph node dissection by bulk excision of tissue including the nodes, enabling a node-to-node comparison between MRI and pathology to validate our nano-MRI results . If successful this technique would form a non-invasive alternative to the current lymph node staging techniques such as surgery. Additionally (if metastatic nodes are present), it could complement image guided focal therapies on lymph node metastases such as radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

General criteria:

* Age > 18 years

Inclusion criteria rectal cancer patients:

* Patients with recently histologically proven rectal cancer, who are planned to undergo a total mesorectal excision without neo-adjuvant radiotherapy.

Inclusion criteria breast cancer patients:

* Patients with recently histologically proven breast cancer (Stage II), who are planned for surgery with sentinel node procedure, but will receive no neo-adjuvant therapy or will undergo an axillary lymph node dissection without prior sentinel node procedure and will receive no neo-adjuvant therapy.

Exclusion Criteria:

General exclusion criteria:

* BMI > 30 kg/m2
* Pregnancy
* Karnofsky score <= 70
* Contraindications for 7T MRI:

  * Epilepsy
  * Inability to provide informed consent
  * Metal implants that are not compatible with 7 Tesla MRI
* Contraindications to USPIO based contrast agents:

  * prior allergic reaction to ferumoxtran-10 or any other iron preparation
  * prior allergic reaction contributed to dextran or other polysaccharide, in any preparation
  * prior allergic reaction to contrast media of any type
  * hereditary hemochromatosis, thalassemia, sickle cell anemia;

Exclusion criteria for rectal cancer:

* Inflammatory diseases of the abdomen (such as Crohn's disease)
* Previous abdominal surgery or radiotherapy

Exclusion criteria for breast cancer:

* Prior radiotherapy or surgery to axillae

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of 7 Tesla MRI in combination with ferumoxtran-10 on nodal level. | within 2 weeks prior to the patients surgery
  The images of the 7 Tesla MRI scan will be evaluated by a radiologist and every lymph node that is found will be scored as positive or negative. This will be compared to the pathological results to determine the sensitivity and specificity of ferumoxtran enhanced MRI on 7 Tesla for diagnosing whether a lymph node is metastatic or not.

SECONDARY OUTCOMES:
Comparison of 7 Tesla and 3 Tesla MRI | within 2 weeks prior to the patients surgery
  The diagnostic accuracy (sensitivity and specificity as described in outcome 1) of 3 Tesla and 7 Tesla will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Tom Scheenen, PhD, Principal Investigator — Radboudumc Nijmegen
Locations (1):
- Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands